CLINICAL TRIAL: NCT05125224
Title: Data Analysis for Drug Repurposing for Effective Alzheimer's Medicines (DREAM)- Dihydropyridine Calcium Channel Blockers Versus Hydrochlorothiazide
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Rutgers University (Other); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Rishi J. Desai, Assistant Professor of Medicine, Brigham and Women's Hospital
Other Study IDs: 2019A010961-6
Record Dates: First submitted 2021-11-08; First posted 2021-11-18 (Actual); Results first posted 2025-11-06 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Hydrochlorothiazide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dihydropyridine calcium channel blocker: Exposure group
  Interventions: Drug: Dihydropyridine calcium channel blocker
- Hydrochlorothiazide: Reference group
  Interventions: Drug: Hydrochlorothiazide

INTERVENTIONS:
Drug: Dihydropyridine calcium channel blocker — Dihydropyridine calcium channel blocker claim is used as the exposure group.
  Groups: Dihydropyridine calcium channel blocker
Drug: Hydrochlorothiazide — Hydrochlorothiazide claim is used as the reference group.
  Groups: Hydrochlorothiazide

SUMMARY:
This study aims to evaluate the comparative risk of dementia/Alzheimer's disease onset between patients treated with medications that target specific metabolic pathways and patients treated with alternative medications for the same indication.

DETAILED DESCRIPTION:
This is a non-randomized, non-interventional study that is part of the DREAM Study of Brigham and Women's Hospital. DREAM is led by Dr. Madhav Thambisetty, MD, PhD, Chief of the Clinical and Translational Neuroscience Section, Laboratory of Behavioral Neuroscience, National Institute on Aging (NIA) intramural research program. This study aims to evaluate the comparative risk of dementia/Alzheimer's disease onset between patients treated with medications that target specific metabolic pathways and patients treated with alternative medications for the same indication using healthcare claims data.

ELIGIBILITY:
Please see https://docs.google.com/spreadsheets/d/1VlyY3zcxoRp0tH7yv8rSOEggSO6WQ0VYEjq-6KlSSt8/edit?usp=sharing or Appendix A for full code and algorithm definitions.

Medicare timeframe: 2008 to 2018 (end of data availability). CRPD timeframe: 2007 to 2018

Inclusion Criteria:

* 1. Aged > 65 years on the index date
* 2. For Medicare - Enrollment in Medicare Part A, B, and D with no HMO coverage for 365 days prior to and including cohort entry date
* 3. At least two claims with hypertension diagnosis recorded in 365 days prior to cohort entry date

Exclusion Criteria:

* 1. Prior history of dementia measured anytime prior to cohort entry date
* 2. Prior use of dihydropyridine CCBs, hydrochlorothiazide, or other antihypertensives anytime prior to cohort entry date

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: This study will employ a new user, active comparator, observational cohort study design comparing dihydropyridine CCBs to hydrochlorothiazide. The patients will be required to have continuous enrollment during the baseline period of 365 days before initiation of dihydropyridine CCBs or hydrochlorothiazide (index date). Follow-up for the outcome (dementia) differs between analyses. Follow-up begins the day after drug initiation (analysis 1, 3, 4); 180 days after drug initiation (analysis 2).
Sampling Method: Non-Probability Sample
Enrollment: 163720 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Madhav Thambisetty, MD, PhD, Principal Investigator — National Institute on Aging (NIA)
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dihydropyridine calcium channel blocker | Hydrochlorothiazide
Started | 77152 | 86568
Completed | 64254 | 64254
Not Completed | 12898 | 22314

BASELINE CHARACTERISTICS:
Population: Medicare - Study cohort after 1:1 propensity score matching
Groups:
- Total: Total of all reporting groups
Arm/Group | Dihydropyridine Calcium Channel Blocker | Hydrochlorothiazide | Total
Number analyzed (Participants) | 64254 | 64254 | 128508
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 64254 | 64254 | 128508
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.44 (6.85) | 73.48 (6.93) | 73.44 (6.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35010 | 34917 | 69927
  Male | 29244 | 29337 | 58581
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 47346 | 47312 | 94658
  Black | 8092 | 8107 | 16199
  Asian | 3295 | 3280 | 6575
  Hispanic | 2463 | 2466 | 4929
  Native American | 471 | 472 | 943
  Other | 1941 | 1962 | 3903
  Unknown | 646 | 655 | 1301
Dementia risk factors [Count of Participants; unit: Participants]
  Diabetes | 45146 | 45024 | 90170
  Obesity | 9833 | 9872 | 19705
  Coronary artery disease | 15043 | 15080 | 30123
  Depression | 7885 | 7906 | 15791
  Anxiety | 7268 | 7252 | 14520
  Bipolar disorder | 747 | 763 | 1510
  Schizophrenia | 468 | 465 | 933

OUTCOME MEASURES:

1. Primary Outcome: Time to Dementia Onset
Description: Time to dementia onset, i.e., Alzheimer's disease, vascular dementia, senile, presenile, or unspecified dementia, or dementia in other diseases classified elsewhere. Please refer to uploaded protocol for full definition due to size limitations.
Time Frame: Median follow up times: 1) 189 days (exp), 171 days (ref) 2) 835 days (exp). 851 days (ref) 3) 388 days (exp), 348 days (ref) 4) 191 days (exp), 172 days (ref)
Measure: Number (95% Confidence Interval); unit: Incidence rate per 1000 person year
Arm/Group | Dihydropyridine calcium channel blocker | Hydrochlorothiazide
Number analyzed (Participants) | 64,254 | 64,254
Incidence rate per 1000 person year
  Analysis 1 | 17.1 [16.2 to 18.0] | 13.7 [12.8 to 14.6]
  Analysis 2 | 20.8 [19.8 to 21.9] | 20.6 [19.6 to 21.6]
  Analysis 3 | 15.6 [14.6 to 16.7] | 13.1 [12.1 to 14.2]
  Analysis 4 | 5.6 [5.1 to 6.2] | 4.0 [3.6 to 4.6]

ADVERSE EVENTS:
Time Frame: 'As-treated' follow-up approach - Median follow-up days of 189 (for Dihydropyridine Calcium Channel Blockers) and 171 (for Hydrochlorothiazide)
Description: Our study did not capture Serious Adverse Events.
Arm/Group | Dihydropyridine calcium channel blocker | Hydrochlorothiazide
All-Cause Mortality (participants affected / at risk) | 0/64254 | 0/64254
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/64254 | 0/64254

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-23): https://cdn.clinicaltrials.gov/large-docs/24/NCT05125224/Prot_SAP_001.pdf